CLINICAL TRIAL: NCT05578807
Title: A Comparative Study of Retrograde Ureteral Catheter Insertion or Not in Total Tubeless Percutaneous Nephrolithotomy
Brief Title: Total Tubeless Percutaneous Nephrolithotomy Without a Ureteral Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Principal Investigator, Li Mingyong, MD, Associate professor, The First Affiliated Hospital of University of South China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020SK51801
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Nephrolithotomy, Percutaneous; Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total tubeless percutaneous nephrolithotomy without reverse insertion of a ureteral catheter (Experimental): In total tubeless percutaneous nephrolithotomy surgery, there is no reverse insertion of a ureteral catheter by transurethral ureteroscopy when a patient is placed in lithotomy position, no need to change the position, and no need to re-sterilize and lay towels.
  Interventions: Procedure: without reverse ureteral catheter insertion
- Conventional total tubeless percutaneous nephrolithotomy (No Intervention): In total tubeless percutaneous nephrolithotomy surgery, there is reverse insertion of a ureteral catheter by transurethral ureteroscopy when a patient is placed in lithotomy position, need to change the position, and need to re-sterilize and lay towels.

INTERVENTIONS:
Procedure: without reverse ureteral catheter insertion — In contrast to conventional total tubeless percutaneous nephrolithotomy, there was no reverse insertion of a ureteral catheter by transurethral ureteroscopy when a patient is placed in lithotomy position, no change in position, and no repeated disinfection.
  Arms: Total tubeless percutaneous nephrolithotomy without reverse insertion of a ureteral catheter

SUMMARY:
Total tubeless Percutaneous nephrolithotomy (PCNL) is a modified surgical method of PCNL surgery, that is, there is no indwelling nephrostomy tube and double-J tube during PCNL surgery. Compared with traditional PCNL surgery, it has the advantages of reducing pain, shortening operation time and reducing operation cost. Since this procedure was first performed in 2004, several randomized clinical studies have verified the safety and efficacy of total tubeless PCNL. Conventional total tubeless PCNL surgery requires the patient to first undergo retrograde transurethral ureteroscopic insertion of the ureteral catheter in the lithotomy position, and then change the patient to the prone position. However, a large number of literature reports and the surgical experience of PCNL in the past 20 years tell the investigators that the reverse insertion of ureteral catheter can cause many recent surgical complications.The study planned to perform the operation in the prone position without reverse insertion of a ureteral catheter in the total tubular PCNL surgery.

DETAILED DESCRIPTION:
The purpose of this single-center, single-blind, randomized trial was to investigate whether without retrograde insertion of a ureteral catheter is appropriate for total tubeless percutaneous nephrolithotomy. It is planned to start in October 2022 and is expected to end in October 2024. Based on inclusion and exclusion criteria, 100 subjects were expected to be recruited. In a parallel group design, subjects were randomly assigned to two groups: the experimental group received total tubeless PCNL without reverse insertion of a ureteral catheter , and the control group received conventional total tubeless PCNL. The primary end point of the study was the incidence of postoperative complications according to the modified Clavien-Dindo complication grading system. Secondary end points included Stone-free rate, operation time, length of hospital stay, and medical costs. Measurement data were expressed as mean ± standard deviation (X ± S), and Student's t-test was used for intergroup comparisons. The counting data were expressed as frequency and percentage, and the chi-squared or Fisher's exact probability test were used for intergroup comparisons. The rank-sum test was used for grade data. P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with kidney stones who met the indications for PCNL surgery.
* the maximum diameter of calculi was less than 35 mm.
* the width of hydronephrosis effusion was less than 25mm.

Exclusion Criteria:

* patients with infectious calculi confirmed by preoperative CT examination and blood biochemical indexes.
* Patients with severe cardiac and pulmonary insufficiency, coagulation dysfunction and other obvious surgical contraindications.
* Patients with previous history of PCNL surgery on the affected side or nephrotomy.
* Patients with indwelling double J tube or nephrostomy tube before operation.
* Patients with renal trauma or congenital anomalies of urinary system.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Rate of fever | From the day of surgery to the day of discharge, up to 2 weeks.
  Fever was defined as axillary temperature greater than 38.5 ° C.
White blood cell count change value | Day 2 before surgery、hour 3 after the surgery
  The change value of White blood cell count between preoperative and
Neutrophils granulocyte change value | Day 2 before surgery、hour 3 after the surgery
  The change value of Neutrophils granulocyte between preoperative and postoperative
Hemoglobin change value | Day 2 before surgery、hour 3 after the surgery
  The change value of Hemoglobin between preoperative and postoperative
Hematocrit change value | Day 2 before surgery、hour 3 after the surgery
  The change value of Hematocrit between preoperative and postoperative
Rate of renal subcapsular hematoma | Day 2 after the surgery
  The proportion of postoperative renal subcapsular hematoma in all patients
Serum creatinine change value | Day 2 before surgery、Hour 3 after the surgery
  The change value of Serum creatinine between preoperative and postoperative
visual analog scale (VAS)pain score | Hour 2 after the surgery
  0: no pain; Less than 3 points: mild pain, tolerable; 4 points to 6 points: the patient's pain and affect sleep, still tolerable; 7-10: Patients have increasing pain, pain is unbearable, affect appetite, affect sleep.
Rate of hydrothorax | Day 2 after the surgery
  Hydrothorax appeared on the surgical side.

SECONDARY OUTCOMES:
Stone free rate | Day 2 after the surgery
  Residual stone less than 4mm in diameter was considered to have been cleared.
Operation time | During the procedure
  Operation time was defined as the time required from the surgeon's handwashing to the completion of surgical incision suture.
length of hospital stay | 2 weeks after surgery
  Length of hospital stay indicated the number of days between the operation date and discharge date
Medical costs | 2 weeks after surgery
  All medical expenses incurred to treat stones.

CONTACTS AND LOCATIONS:
Overall Officials: Mingyong Li, MD., Study Director — the First Affiliated Hospital of the University of South China
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to other researchers after the study Report are published.
Supporting Information: Study Protocol, ICF
Time Frame: One year after the study report was published,but the duration is uncertain.
Access Criteria: When proper editing or review requirements are met, the study data will be available from the study manager after the study is completed.

DOCUMENTS (1):
  • Study Protocol (2022-10-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT05578807/Prot_000.pdf